CLINICAL TRIAL: NCT01276496
Title: A Phase I, Open Label, Dose Escalation Study of the Safety, Tolerability and Pharmacokinetic Properties of the Combination of Cilengitide and Paclitaxel in Patients With Advanced Solid Malignancies
Brief Title: Weekly Doses of Cilengitide and Paclitaxel in Treating Patients With Advanced Solid Tumors That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00619; NCI-2013-00619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01CA069912 (NIH); MC0915 (Other: Mayo Clinic); 8335 (Other: CTEP); P30CA015083 (NIH); NCT01647139 (obsolete NCT alias)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2015-03

CONDITIONS: Adult Solid Neoplasm; Estrogen Receptor Negative; HER2/Neu Negative; Male Breast Carcinoma; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Cilengitide; Paclitaxel; Taxes

ARMS (1):
- Treatment (cilengitide, paclitaxel) (Experimental): Patients receive cilengitide IV over 1 hour on days* 1, 8, and 15 and paclitaxel IV over 1 hour on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  NOTE: *Some patients receive cilengitide IV over 1 hour on days 1, 2, 8, 9, 15, and 16.
  Interventions: Drug: Cilengitide; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cilengitide — Given IV
  Other Names: EMD 121974; EMD-121974
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of cilengitide when given together with paclitaxel weekly in treating patients with solid tumors that have spread nearby or to other areas of the body and cannot be removed by surgery. Cilengitide may stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel, work in different ways to the stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cilengitide together with paclitaxel may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) of cilengitide and paclitaxel at weekly dose schedule. (Cohort I) II. To describe the toxicities associated with cilengitide and paclitaxel. III. To describe any antitumor activity of cilengitide and paclitaxel at weekly dose schedule.

IV. To characterize pharmacokinetics (PK) of cilengitide and paclitaxel with the proposed schedule and correlate PK parameters to clinical outcome. (Cohort I) V. To examine the effect of cilengitide and paclitaxel on circulating cysteine-rich, angiogenic inducer, 61 (Cyr61) using a novel "sandwich enzyme-linked immunosorbent assay (ELISA)" and to correlate this effect with clinical response. (Cohort II) VI. To evaluate the information obtained through use of items from the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) in Phase I studies.

VII. To determine if tumor tissue expression of alpha v beta 3 (αvβ3) and CYR61 correlate with therapeutic response to cilengitide with paclitaxel. (Cohort II)

OUTLINE: This is a dose-escalation study of cilengitide.

Patients receive cilengitide intravenously (IV) over 1 hour on days* 1, 8, and 15 and paclitaxel IV over 1 hour on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Some patients receive cilengitide IV over 1 hour on days 1, 2, 8, 9, 15, and 16.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer that is now unresectable (solid tumors, excluding lymphoma)
* For Cohort II only:

  * Histologic adenocarcinoma of the breast with manifestations of metastatic cancer or locally advanced, unresectable cancer
  * Estrogen, progesterone, and human epidermal growth factor receptor 2 (HER2) receptor negative disease per local standards
  * Refractory to taxanes which is defined as one of the following:
  * Having relapsed during or within 12 months of completing adjuvant paclitaxel or docetaxel
  * Disease progression while on any taxane in the locally advanced, unresectable or metastatic breast cancer setting
  * Ability and willingness to undergo biopsy for biomarker testing prior to start of treatment
  * Disease must be measurable by imaging-based evaluation per Response Evaluation Criteria in Solid Tumors (RECIST) criteria (v1.1)
  * Up to 5 prior regimens of chemotherapy for metastatic disease are allowed
* Absolute neutrophil count (ANC) >= 1500/μL
* Hemoglobin (Hgb) >= 9 g/dL
* Platelets (PLT) >= 100,000/μL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 3 x ULN or AST =< 5 x ULN if liver involvement
* Creatinine =< 1.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, or 1 (or Karnofsky performance status [KPS] > 70)
* Ability to provide informed consent
* Willingness to return to the enrolling Mayo Clinic institution for follow-up
* Life expectancy >= 12 weeks
* All patients: Willingness to provide blood samples for the mandatory correlative research component
* For Cohort II, tissue biopsies are mandatory
* Women of childbearing potential only: negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential including women within 2 years of post-menopause

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy =< 21 days prior to registration
  * Mitomycin C/nitrosoureas =< 42 days prior to registration
  * Immunotherapy =< 14 days prior to registration
  * Biologic therapy =< 14 days prior to registration
  * Prior investigational therapy =< 28 days prior to registration
  * Full field radiation therapy =< 28 days prior to registration or limited field radiation therapy < 14 days prior to registration

    * Full field radiation encompasses the entire area of known disease involvement and surrounding uninvolved but at-risk areas, e.g. subtotal nodal (mantle and upper abdomen) or total nodal irradiation
    * Limited field radiation is restricted to treating only the known areas of clinical disease, e.g. involved-field therapy for lymphoma
  * Major surgery (i.e., laparotomy) =< 4 weeks prior to registration; minor surgery =< 2 weeks prior to registration; Note: insertion of a vascular access device is not considered major or minor surgery in this regard
* Unresolved toxicities from prior therapy with the exception of alopecia that have not resolved to =< grade 1, unless the patient has a chronic, stable =< grade 2 toxicity that would not interfere with the evaluation of the study agents
* New York Heart Association classification III or IV
* Central nervous system (CNS) metastases or seizure disorder; Note: CNS metastases are allowed if previously treated and stable for at least 4 weeks
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragm, injections, intrauterine device [IUD], or abstinence, etc.); oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive on highly active antiretroviral therapy (HAART) therapy
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: nonmelanotic skin cancer or carcinoma-in-situ of the cervix; Note: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Uncontrolled hypertension, labile hypertension of history of poor compliance with antihypertensive medication
* Patients with active, bleeding diathesis
* Non-disease related- major surgery, =< 28 days or minor surgery =< 7 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Best response, defined to be complete response (CR) or partial response (PR) as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | From start of the treatment until disease progression/recurrence, assessed up to 3 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Change in Cyr61 expression levels (Cohort II) | Baseline to up to 3 months
  At the end of each cycle, the percent change in serum Cyr61 expression from pre-treatment levels will be determined for each patient. For each patient, a times series plot of the percent change in serum Cyr61 expression from pre-treatment levels will be constructed and visually inspected for trends across time as well as for differences between those who respond to treatment (CR or PR by RECIST criteria) and those who do not.
Change in Cyr61 expression levels (Cohort II) | Baseline to 21 days
  A Wilcoxon rank sum test will be used to assess the percent change in Cyr61expression level after one cycle of treatment from pretreatment levels differs between those who progress within 120 days (within the first 6 cycles of treatment) and those who remain progression-free at least 120 days.
Incidence of grade 3+ adverse events, as graded using NCI CTCAE v 4.0 | Up to 3 months
  The number and severity of grade 3+ adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population.
Incidence of hematologic toxicity, including thrombocytopenia, neutropenia, and leukopenia, evaluated via the ordinal CTC | Up to 3 months
  Assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Incidence of non-hematologic toxicity, evaluated via the ordinal Common Toxicity Criteria (CTC) | Up to 3 months
  Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
MTD of cilengitide and paclitaxel, defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least 1/3 of patients as graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | 3 weeks
Number of all adverse events, graded according to the NCI CTCAE v4.0 | Up to 3 months
  The number of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population.
Overall survival (OS) (Cohort II) | The time of registration to death due to any cause, assessed up to 3 months
  Kaplan-Meier method will be used to estimate the distribution of OS time.
Progression-free survival (PFS) (Cohort II) | The time of registration to documentation of disease event where a disease event is local/regional/distant progression, contralateral breast disease, second primary disease or death due to any cause, assessed up to 3 months
  Kaplan-Meier method will be used to estimate the distribution of PFS time.
Response rate, defined as the proportion of patients whose tumor responds to treatment (Cohort II) | Up to 3 months
  Calculated as the number of eligible patients whose tumor meets the criteria for a CR or PR on two consecutive evaluations at least 6 weeks apart divided by the number of eligible patients with metastatic breast cancer refractory to taxanes who begin treatment. A 95% binomial confidence interval will be constructed for the true response rate.
Severity of all adverse events, graded according to NCI CTCAE v4.0 | Up to 3 months
  The severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population.
Time to progression | Up to 3 months
Time to treatment failure | Time from registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months
Time until any treatment related toxicity | Up to 3 months
Time until hematologic nadir for ANC | Up to 3 months
Time until hematologic nadir for platelets | Up to 3 months
Time until hematologic nadir for WBC | Up to 3 months
Time until treatment related grade 3+ toxicity | Up to 3 months

SECONDARY OUTCOMES:
Incidence of toxicity, as assessed using PRO-CTCAE | Up to 3 months
  The PRO-CTCAE will be summarized descriptively, and the dropout rate will be used for feasibility study. Informal comparison and correlation of the PRO-CTCAE symptoms with their corresponding items in clinician reported CTCAE will be conducted in an exploratory manner. Chi-squared tests will be used without adjustment for multiple comparisons.

OTHER OUTCOMES:
Pharmacokinetic (PK) parameters of cilengitide, including area under curve (AUC), maximum concentration Cmax and trough plasma concentrations | Baseline; 1, 1.5, 2, 3, 4, and 5 hours post-cilengitide day 1 of courses 1 and 2; 27 hours post-paclitaxel day 2 of courses 1 and 2
  Analyses will be primarily descriptive in nature. PK parameters will be determined from the individual plasma concentration-time curves of cilengitide, using non-compartmental and/or compartmental models. These parameters will be correlated to clinical outcomes such as tumor response. The possible effects of cilengitide upon paclitaxel pharmacokinetics, and vice-versa, will be explored using standard parametric or non-parametric techniques.
PK parameters of paclitaxel, including AUC, Cmax and trough plasma concentrations | Baseline; 1, 1.5, 2, 3, 4, and 5 hours post-cilengitide day 1 of courses 1 and 2; 27 hours post-paclitaxel day 2 of courses 1 and 2
  Analyses will be primarily descriptive in nature. PK parameters will be determined from the individual plasma concentration-time curves of paclitaxel, using non-compartmental and/or compartmental models. These parameters will be correlated to clinical outcomes such as tumor response. The possible effects of cilengitide upon paclitaxel pharmacokinetics, and vice-versa, will be explored using standard parametric or non-parametric techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Molina, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota